CLINICAL TRIAL: NCT06436729
Title: Impact of MINST With and Without Splinting on Clinical Periodontal Parameters and OHRQoL in Periodontitis Patients With Mobile Anterior Teeth: A Randomized Controlled Trial
Brief Title: Impact of MINST With and Without Splinting in Periodontitis Patients With Mobile Anterior Teeth
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Navi Bansal Perio 24/39
Record Dates: First submitted 2024-05-24; First posted 2024-05-31 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Tooth Mobility; Periodontitis
Keywords: Splinting; OHRQoL; MINST
MeSH Terms: conditions — Tooth Mobility; Periodontitis | interventions — Splints

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MINST with Splinting (Experimental): Minimally Invasive Non-Surgical Therapy will be done along with splinting of mobile anterior teeth
  Interventions: Procedure: Splinting
- MINST without Splinting (Active Comparator): Minimally Invasive Non-Surgical Therapy will be done without splinting of mobile anterior teeth
  Interventions: Procedure: MINST alone

INTERVENTIONS:
Procedure: Splinting — The joining of two or more teeth into a rigid unit by means of a fixed or removable restorations/devices
  Arms: MINST with Splinting
Procedure: MINST alone — Minimally invasive non surgical therapy alone
  Arms: MINST without Splinting

SUMMARY:
The goal of this clinical trial is to evaluate impact of Minimally Invasive Non-Surgical Therapy (MINST) with and without splinting on clinical periodontal parameters and Oral Health Related Quality of Life (OHRQoL) in periodontitis patients with mobile anterior teeth. The main questions it aims to answer are:

* Does splinting provide additional benefit to MINST alone for improving the clinical periodontal parameters ?
* Does splinting provide additional benefit to MINST alone for improving OHRQoL ?

DETAILED DESCRIPTION:
The increased mobility of a periodontally affected tooth can be caused by a shift of centre of rotation of the tooth apically due to clinical attachment loss (CAL) and alveolar bone loss (ABL) and/or due to secondary occlusal trauma.

Tooth splinting continues to be a topic of controversy. It remains one of the most poorly understood and controversial areas of dental therapy.

Minimally invasive non-surgical periodontal therapy (MINST) has been introduced for minimizing tissue trauma and enhancing clinical outcomes by the adjunctive use of magnification devices .

This study aims to compare clinical periodontal parameters and Oral Health Related Quality of Life (OHRQoL) following Minimally Invasive Non-Surgical Therapy (MINST), both with and without splinting, in patients with Stage III and Stage IV periodontitis who have mobile anterior teeth.

Patients will be screened and enrolled based on specific eligibility criteria. Baseline measurements of outcome parameters will be taken, followed by supragingival scaling, and patients will be recalled after one week.

During the subsequent visit, patients will be randomized into either the test group or the control group. The test group will receive MINST along with splinting of the mobile anterior teeth, while the control group will receive MINST alone.

Patients will be recalled after 8 weeks and 6 months to assess changes in the outcome measurements.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria at the patient level: systemically healthy patient with presence of stage III or IV periodontitis, age ≥ 18 years.
* Tooth-related inclusion criteria: presence of at least one anterior tooth with mobility in combination with a clinical attachment loss (CAL) ≥ 5 mm and a relative alveolar bone loss (ABL) of ≥ 50% at the affected tooth.
* Dentition with at least 3 antagonistic contact zones opposing posterior teeth, that is Eichner Class A1, A2, A3, B1

Exclusion Criteria:

* Patients with anterior cross bite
* Bruxism or signs of parafunction
* Implant in Anterior teeth
* Any active periodontal therapy in last 1 year
* Mobility of teeth due to acute trauma
* Pulpal or periapical pathology in anterior teeth
* Patient requiring any emergency dental procedure
* Patient on antibiotic therapy in last 1 month
* If patient want to undergo surgical treatment for management of periodontitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Clinical Attachment Level (CAL) | 12 - 14 months
  Clinical attachment level is the distance between the cemento-enamel junction and the base of pocket.
Changes in Oral Health Related Quality of Life (OHRQoL) | 12 - 14 months
  OHRQoL will be measured using a validated version of Oral Health Index Profile (OHIP)

CONTACTS AND LOCATIONS:
Overall Officials: Navi Bansal, BDS, Principal Investigator — PGIDS, ROHTAK
Locations (1):
- PGIDS, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: No